CLINICAL TRIAL: NCT06417970
Title: The Relationship Between Shoulder Proprioception, Palmar Touch Sensation and Psychometric Parameters in Volleyball Players
Brief Title: Proprioception, Touch and Psychometric Relationship in Volleyball Players
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Ramazan Kursat Erdas, Dr, Suleyman Demirel University
Other Study IDs: Voleybolcu Omuz
Record Dates: First submitted 2024-04-23; First posted 2024-05-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Proprioceptive Disorders; Sports Physical Therapy; Kinesiophobia; Somatosensory Disorders; Shoulder Injuries
MeSH Terms: conditions — Somatosensory Disorders; Kinesiophobia; Shoulder Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Volleyball Players
  Interventions: Diagnostic Test: Shoulder Proprioception, Palmar Touch Sensation and Psychometric Parameters

INTERVENTIONS:
Diagnostic Test: Shoulder Proprioception, Palmar Touch Sensation and Psychometric Parameters — Shoulder Proprioception: Proprioception will be measured with isokinetic device. The measurement reference angles are 30° and 60°.
  Palmar Touch Sensation: Palmar tactile sensation will be measured with the Semmes-Weinstein Monofilament.
  Psychometric Parameters: Athlete Psychological Strain Questionnaire, Tampa kinesiophobia questionnaire

SUMMARY:
Improvement of proprioception in athletes has been found to be effective in preventing fear of movement. The importance of these parameters has not been sufficiently emphasized in volleyball players. In addition, the relationship between upper extremity proprioception and the sense of touch, which is an important component of the somatosensory system, and common anxiety states in athletes has not been evaluated. Therefore, the aim of our study was to investigate the relationship between shoulder joint proprioception and psychometric parameters, kinesiophobia and palmar tactile sensation in volleyball players.

DETAILED DESCRIPTION:
The study will not include any intervention program. Volleyball players who are volleyball players in their school team and volleyball players who apply to the Sports Medicine Polyclinic with a general health examination or lower extremity injury complaint will be invited to the study. Volleyball players between the ages of 18-30, who meet the inclusion criteria and consent to participate will be included in the study. At the beginning, the participants will be informed and if they volunteer, they will sign an informed consent form. The demographic data of the participants will be filled in on a form prepared by the researchers.

The parameters to be evaluated during the study are glenohumeral joint proprioception measurements (internal rotation, external rotation), Athlete Psychological Strain Questionnaire, Tampa Kinesiophobia Questionnaire and palmar tactile sensation measurement with Semmes-Weinstein Monofilament.

Glenohumeral joint proprioception measurements: Visual input is eliminated with a blindfold while the participant is in a seated position with the arm in 90° abduction and elbow in 90° flexion. The measurement reference angles are 30° and 60°. The upper extremity will be moved passively from the neutral position in the direction of internal and external rotation up to the reference angle. It will be held at the reference angle for 10 seconds and then passively moved back to the neutral position. The speed of the dynamometer will be set to 0.5°/s. The participant will then be instructed to repeat the position in which the upper limb was previously placed, taking into account the reference angle. After the learning trial, the average of the absolute error of the three test trials will be recorded as the position sense test result.

Athlete Psychological Strain Questionnaire: This questionnaire will be used to measure sport-specific psychological tension. It consists of 10 items and each item is scored on a 5-point Likert scale (1=never to 5=always) and assesses self-regulation (e.g. "I felt less motivated"), performance (e.g. "I found training more stressful") and external coping (e.g. "I took unusual risks off the field"). The minimum score is 10, while the maximum score is 50. Higher scores indicate greater psychological strain.

Tampa kinesiophobia questionnaire: This questionnaire measures fear of movement/reinjury. It consists of 17 items and the normal score range is between 17 and 68. A lower score indicates a better condition.

Palmar tactile sensation: Palmar tactile sensation will be measured with the Semmes-Weinstein Monofilament. The tested hand will be placed on a towel and hidden behind a screen with the forearm supinated. Monofilaments will be placed in contact with the tip of the thumb (median nerve), the tip of the little finger (ulnar nerve) and between the index finger and thumb on the dorsal side of the hand (radial nerve). Patients will be asked to verbally answer "Yes" when they feel touched by the monofilaments. The monofilament will be applied perpendicular to the skin until it is slightly bent for 1.5 seconds. The measurement time (approach, pressure and withdrawal of the monofilament) will not exceed 3 seconds and the test will start with the thinnest monofilament (lowest pressure) and end when at least 1 positive response is collected from 3 trials.

The power analysis of the study was performed with the program GPower 3.1.9.7 (Universitaet Kiel, Germany). In the study, the correlation value between the Y-Balance Test Inferolateral and Internal Rotation Active Joint Position Sensation measurements calculated in Mendez-Rebolledo et al. (2022), r=-0.57, was used. Accordingly, test family "Exact" and analysis type "Correlation: Bivariate normal model" were selected. The explanatory coefficient R2=0.33 and the alternative hypothesis effect size was calculated as 0.574. The sample size was determined as n=33 with a two-way table value, 95% power and 5% type-I margin of error.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-30 years old
* Being a sub-elite level volleyball player (school team / student athlete)
* Regular volleyball training (at least once a week)
* No history of upper extremity injury in the last 1 year

Exclusion Criteria:

* Having undergone a surgery involving the upper extremity
* Any orthopedic problems that may affect the assessments
* Not giving consent to participate in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volleyball athlete
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Glenohumeral joint proprioception measurement | Change from Baseline glenohumeral joint proprioception measurement at first day
  Visual input is eliminated with a blindfold while the participant is in a seated position with the arm in 90° abduction and elbow in 90° flexion. The measurement reference angles are 30° and 60°. The upper extremity will be moved passively from the neutral position in the direction of internal and external rotation up to the reference angle. It will be held at the reference angle for 10 seconds and then passively moved back to the neutral position. The speed of the dynamometer will be set to 0.5°/s. The participant will then be instructed to repeat the position in which the upper limb was previously placed, taking into account the reference angle. After the learning trial, the average of the absolute error of the three test trials will be recorded as the position sense test result.
Athlete Psychological Strain Questionnaire | Change from Baseline Athlete Psychological Strain Questionnaire at first day
  This questionnaire will be used to measure sport-specific psychological tension. It consists of 10 items and each item is scored on a 5-point Likert scale (1=never to 5=always) and assesses self-regulation (e.g. "I felt less motivated"), performance (e.g. "I found training more stressful") and external coping (e.g. "I took unusual risks off the field"). The minimum score is 10, while the maximum score is 50. Higher scores indicate greater psychological strain.
Tampa kinesiophobia questionnaire | Change from Baseline Tampa kinesiophobia questionnaire at first day
  This questionnaire measures fear of movement/reinjury. It consists of 17 items and the normal score range is between 17 and 68. A lower score indicates a better condition.
Palmar tactile sensation | Change from Baseline palmar tactile sensation at first day
  Palmar tactile sensation will be measured with the Semmes-Weinstein Monofilament. The tested hand will be placed on a towel and hidden behind a screen with the forearm supinated. Monofilaments will be placed in contact with the tip of the thumb (median nerve), the tip of the little finger (ulnar nerve) and between the index finger and thumb on the dorsal side of the hand (radial nerve). Patients will be asked to verbally answer "Yes" when they feel touched by the monofilaments. The monofilament will be applied perpendicular to the skin until it is slightly bent for 1.5 seconds. The measurement time (approach, pressure and withdrawal of the monofilament) will not exceed 3 seconds and the test will start with the thinnest monofilament (lowest pressure) and end when at least 1 positive response is collected from 3 trials.

SECONDARY OUTCOMES:
Demographic data | Change from Baseline demographic data at first day
  Whether the athlete is healthy or not, age, gender, height, weight, history of upper extremity injuries, presence of chronic diseases, sport position, weekly training frequency, how long he/she has been playing volleyball, dominant side, shoulder range of motion will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ferdi Başkurt, PhD, Principal Investigator — Süleyman Demirel University; Sabriye Ercan, PhD, Study Director — Süleyman Demirel University; Elif Şahin, MSc, Study Chair — Süleyman Demirel University; İsmet Tümtürk, MSc, Study Chair — Süleyman Demirel University; Ramazan Kürşat Erdaş, MD, Study Chair — Süleyman Demirel University; Fatih Uğur Taş, MD, Study Chair — Süleyman Demirel University; Furkan Hasan Küçük, MD, Study Chair — Süleyman Demirel University
Locations (1):
- Süleyman Demirel University Faculty of Medicine, Clinic of Sports Medicine, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No